CLINICAL TRIAL: NCT05363020
Title: S-Adenosyl-L-Methionine (SAMe) vs Placebo for Discomfort and Functional Limitations Associated With Osteoarthritis of the Hands: a Pilot Study
Brief Title: S-Asenosyl-L-Methionine vs Placebo for Osteoarthritis of the Hands
Acronym: SAMe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Scott C. Jaynes, Physician Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY02001354
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis Hand
Keywords: SAMe; S-Adenosyl-L-Methionine
MeSH Terms: interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-Adenosyl-L-Methionine (SAMe) (Experimental): Participants receive S-Adenosyl-L-Methionine (SAMe) 400mg capsule orally twice daily for 8 weeks, followed by a 1 week washout period.
  Interventions: Drug: S-Adenosyl-L-Methionine (Sam-E); Drug: Placebo
- Placebo (Placebo Comparator): Participants receive identically appearing 400mg capsule orally twice daily for 8 weeks, followed by a 1 week washout period.
  Interventions: Drug: S-Adenosyl-L-Methionine (Sam-E); Drug: Placebo

INTERVENTIONS:
Drug: S-Adenosyl-L-Methionine (Sam-E) — 400 mg capsule
Drug: Placebo — 400 mg identically appearing placebo

SUMMARY:
The primary objective of this study is to demonstrate the feasibility of evaluating SAMe tolerability, analgesic benefits, and daily functional improvement in patients with osteoarthritis of the hands compared to placebo. The secondary objective of this study is to generate preliminary data on discomfort, function, quality of life in patients with osteoarthritis of the hands when taking SAMe compared to placebo.

DETAILED DESCRIPTION:
At week 0, all patients giving written informed consent and meeting eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to SAMe (400mg orally, twice daily) or placebo (400mg, twice daily) for 8 weeks. Followed by a one week wash out period followed by another 8 weeks of SAMe (400mg, twice daily) or placebo (400mg, twice daily) for 8 weeks (whichever was not given during the first 8 week period).

Participants will complete weekly surveys during the entire study regarding hand discomfort, functional limitations and side effects

ELIGIBILITY:
Inclusion Criteria:

* Current primary care provider within the Dartmouth Health system
* Office visit at Dartmouth Health in the past 3 years
* Participants must be 40 or older at the time of signing the informed consent
* Participants have discomfort or functional limitations of one or both hands AND either:

  1. Objective findings of at least one hand meeting diagnostic criteria based on the American College of Rheumatology (ACR)* or
  2. Existing radiographic evidence of osteoarthritis as judged by a radiologist
* Patients taking OTC or prescription analgesics who are willing to stop their current analgesics for two weeks prior to study entry and remain off those medications over the course of the study
* *Objective inclusion criteria (see poster schematic)

Swelling or deformity of 2 of the following ten joints: the 2nd and 3rd distal interphalangeal (DIP) of each hand, the 2nd and 3rd proximal interphalangeal (PIP) of each hand, and the 1st carpometacarpal joints of both hands.

Exclusion Criteria:

* Patients taking prescription medications other than NSAIDs for their OA who are unable to stop their medication
* Patients with diagnoses of arthritis from conditions other than OA
* Patients whose symptomatic joint is an artificial joint
* Patients with Bipolar Disorder
* Patients taking any of the following medications at study entry OR starting any of these medications during the study period:

  1. daily opioids (including tramadol or buprenorphine)
  2. gabapentin or pregabalin
  3. prednisone
  4. Prescription NSAIDs that they are unable to stop or topical diclofenac
  5. SNRI drugs (Effexor, Cymbalta, Fetzima, Pristiq)
* The participant has a condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Determine the effect of SAMe supplements on hand discomfort relative to placebo, as measured by the change in discomfort scores over time on a visual analog scale | Weekly for 17 weeks
  Scores range from 0-10, 0 being no discomfort and 10 being maximum discomfort

SECONDARY OUTCOMES:
Determine the effect of SAMe supplementation on quality of life measures regarding hand arthritis, as measured by DASH (Disability of Arm, Shoulder and Hand) survey responses done weekly for 17 weeks | Weekly for 17 weeks
  Survey using descriptors of disability and function ranging from no disability to complete disability with 3 other levels of disability in between done weekly for 17 weeks
Determine tolerability of SAMe supplementation compared to placebo, as measured by a survey of 14 common symptoms one may experience from a supplement | Weekly for 17 weeks
  14 symptoms queried for occurrence over the week ranging from "Not at All" to "Very Much" with three additional options in between

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Jaynes, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No